CLINICAL TRIAL: NCT00197704
Title: Nutrition, Immunology and Epidemiology of Tuberculosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Muhimbili University of Health and Allied Sciences (Other)
Responsible Party: Wafaie Fawzi, Harvard School of Public Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AI45441
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2010-11-11 (Estimated); Status verified 2010-11

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; HIV; Tanzania; multivitamins
MeSH Terms: conditions — Tuberculosis | interventions — Geritol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo
- Multivitamins (Experimental): 5000 IU of retinol, 20 mg of B1, 20 mg of B2, 25 mg of B6, 100 mg of niacin, 50 mcg of B12, 500 of C, 200 mg of E, 0.8 mg of folic acid, and 100 mcg of selenium
  Interventions: Dietary Supplement: Multivitamins

INTERVENTIONS:
Dietary Supplement: Multivitamins — 5000 IU of retinol, 20 mg of B1, 20 mg of B2, 25 mg of B6, 100 mg of niacin, 50 mcg of B12, 500 of C, 200 mg of E, 0.8 mg of folic acid, and 100 mcg of selenium taken orally on a daily basis from the start of TB therapy through 8 months of anti-TB therapy
  Arms: Multivitamins
Other: Placebo — Placebo pill taken orally on a daily basis from the start of TB therapy through 8 months of anti-TB therapy
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy of micronutrient supplementation among patients with active tuberculosis, half of who are co-infected with HIV-1

DETAILED DESCRIPTION:
Tuberculosis (TB) remains the single most common infectious disease cause of mortality. We propose to examine the inter- relationships of nutrition, immunology, and epidemiology with respect to TB in Tanzania. Given that TB is so much linked with HIV immunologically, clinically, and epidemiologically, it is essential to examine how these relationships are modified by HIV infection. Published animal and human studies suggest that vitamin deficiency is associated with poor immune response in TB. By modulating immune function, nutritional supplements may be a useful adjunct to anti-TB drugs, and could lead to the development of shorter drug regimens. All patients will receive standard anti-TB therapy. Follow-up visits will occur every two weeks for the first 2 months and monthly thereafter till the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age 18 to 60 years inclusive
* At least two positive sputum smears for tuberculosis
* Intention to stay in Dar-es-Salaam for at least 2 years after the start of TB therapy
* Subjects who grant informed consent to participation

Exclusion Criteria:

* Karnofsky score < 40%
* Hemoglobin < 8.5 g/dl
* Having had treatment for TB exceeding 4 weeks in the last 5 years
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 876 (Actual)
Dates: Start 2000-03; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy of micronutrient supplements on sputum conversion, survival, and TB relapse and reinfection. | Sputum and culture negativity: 1 month and 2 months; Survival: 8 months and 24 months; TB relapse and reinfection: throughout follow-up.

SECONDARY OUTCOMES:
To examine the effect of micronutrient supplements on HIV viral load, CD4 counts, body weight and immunological parameters. | Rate of change of HIV viral load in HIV positive patients: 2, 5, 8, and 20 months; Absolute change in CD4 counts: 2, 5, 8, and 20 months; Weight change from baseline: 2, 8, and 20 months; Immunological parameters: 2, 8, and 20 months.

CONTACTS AND LOCATIONS:
Overall Officials: Wafaie W Fawzi, MD,DrPh, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Harvard School of Public Health, Boston, Massachusetts, United States

REFERENCES:
- [Result] Villamor E, Mugusi F, Urassa W, Bosch RJ, Saathoff E, Matsumoto K, Meydani SN, Fawzi WW. A trial of the effect of micronutrient supplementation on treatment outcome, T cell counts, morbidity, and mortality in adults with pulmonary tuberculosis. J Infect Dis. 2008 Jun 1;197(11):1499-505. doi: 10.1086/587846. PMID 18471061
- [Derived] Mehta S, Mugusi FM, Bosch RJ, Aboud S, Urassa W, Villamor E, Fawzi WW. Vitamin D status and TB treatment outcomes in adult patients in Tanzania: a cohort study. BMJ Open. 2013 Nov 18;3(11):e003703. doi: 10.1136/bmjopen-2013-003703. PMID 24247327